CLINICAL TRIAL: NCT05476640
Title: The Application of Targeted Sequencing in the Screening of Neonatal Diseases
Brief Title: Newborn Sequencing Screening in China
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Children's Hospital (Other)
Collaborators: Children's Hospital of Chongqing Medical University (Other); Xuzhou maternal and Child Health Care Hospital (Unknown); Northwest Women's and Children's Hospital, Xi'an, Shaanxi (Other); Zunyi Maternal and Child Health Care Hospital (Unknown); Inner Mongolia Maternal and Child Health Care Hospital (Other); Huzhou Maternity and Child Health Care Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: shercru-20220003
Record Dates: First submitted 2022-07-19; First posted 2022-07-27 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Newborns

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A dry blood spot was made on the basis of routine blood collection.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- National multicenter screening: NGS was performed based on conventional NBS. The relationship between NGS detected gene variation and disease occurrence was studied through follow-up.
  Interventions: Genetic: NGS

INTERVENTIONS:
Genetic: NGS — In the Nation multicenter screening cohort, NGS testing was performed on the basis of conventional NBS to study the relationship between gene variation and disease occurrence;

SUMMARY:
The project will carry out the genetic testing of 10000 neonates. The aim of the project is to assess the application of targeted sequencing technology in the screening of neonatal diseases.

DETAILED DESCRIPTION:
Neonatal screening (NBS) is the last step of birth defects prevention. Currently, biochemical and mass spectrometry are commonly used for NBS, but there are limited diseases and certain false positive/negative. High-throughput sequencing (NGS) has been widely used in prenatal diagnosis, tumor-targeted biomarkers detection and pathogen detection. Although the application of NGS in new screening has a broad prospect and many countries around the world have begun to explore it, there are still challenges in the selection of screening diseases, gene clinical phenotypes, genetic counseling and clinical pathway.

Since 2019, our team began to explore the appllication of NGS technologies in the clinical application of tertiary prevention, combined with Clinva, HGMD, OMIM database, on the basis of screening specific disease-causing genes and mutation sites as the target, A NGS panel for Newborns in China (NeoExome) was designed, covering 542 single-gene diseases with 601 genes. The rationality and validity of the NGS panel was preliminarily verified in 3423 neonatal blood samples collected from 5 new screening centers in China.

In order to further optimize the gene screening spectrum of neonatal diseases in the Chinese population, evaluate the efficacy of targeted sequencing technology in the screening and diagnosis of neonatal diseases, standardize the clinical pathway, and lay a foundation for the formulation of China's new screening NGS guidelines, the investigators further optimized the targeted sequencing package (NeoexOME-V2) on the basis of the first phase. 491 genes covering 485 single-gene genetic diseases were designed to launch the "Budding Action". The project plans to collect 10000 samples nationwide and carry out the multi-center clinical research on the application of targeted sequencing technology in the screening of neonatal diseases.

ELIGIBILITY:
Inclusion Criteria:

* -- Subjects: all newborns (from birth to 28 days);
* -- After fully understanding the program, the guardian signs the informed consent and agrees to participate in the program.

Exclusion Criteria:

* Other similar clinical research projects are under way for the examined neonates;
* Neonates have received transfusion of allogeneic blood products;
* Newborns whose guardians explicitly refuse to participate in the program after receiving the mission.

Elimination criteria

* Samples that are not properly collected or stored for testing;
* Samples with non-standard data records;
* Samples without clinical follow-up results;
* The project recalls newborns who are required to withdraw by their guardians during the follow-up.

Ages: 1 Day to 28 Days | Sex: All
Age Groups: Child
Study Population: All newborns are our targeted population.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2022-08-05 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease incidence among NGS positive participants | 3 years
  Newborn was followed up for 3 years after birth, and the follow-up results were compared to evaluate and study the relationship between gene variation and disease occurrence

SECONDARY OUTCOMES:
The consistency of test results of NGS and conventional NBS | 1 year
  Conventional NBS was used as the standard to study the application potential of targeted sequencing technology in neonatal screening and evaluate its consistency

CONTACTS AND LOCATIONS:
Overall Officials: Lin Zou, Principal Investigator — Shanghai Children's Hospital

IPD SHARING:
Plan to Share IPD: Undecided